CLINICAL TRIAL: NCT05312710
Title: Phase 2 Study to Evaluate the Safety and Efficacy of APG-157 as Neoadjuvant/Induction Therapy for Patients With Head and Neck Squamous Cell Cancer (HNSCC) of the Oral Cavity and/or Oropharynx
Brief Title: Safety and Efficacy of APG-157 in Head and Neck Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aveta Biomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVTA 20-01
Record Dates: First submitted 2022-03-16; First posted 2022-04-05 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma of Oral Cavity; Squamous Cell Carcinoma of the Oropharynx
Keywords: Neoadjuvant; Induction Therapy; Oral Cancer; Oropharyngeal Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms; Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APG-157 (Experimental): Two pastilles (100 mg) taken three times a day (i.e. before meal time).
  Interventions: Drug: APG-157

INTERVENTIONS:
Drug: APG-157 — Treatment

SUMMARY:
The purpose of this clinical research study is to study safety and efficacy of orally administered APG-157 as the neoadjuvant/induction therapy in newly diagnosed, locally advanced patients with Head & Neck Cancer of oral cavity and/or oropharynx.

The study hypothesis is that neoadjuvant use of APG-157 will reduce the tumor burden prior to any definitive therapy to improve the outcomes over current standard of care.

DETAILED DESCRIPTION:
The patient will receive neoadjuvant therapy (APG-157) during the period between initial diagnosis and time of definitive treatment. APG-157 is an orally administered drug in a form of pastille (soft lozenge) taken three times a day. It dissolves in the mouth. After the neoadjuvant treatment, the patient undergoes surgery or any other definitive therapy and/or postoperative radiotherapy as determined by the patient's doctor. Duration of treatment is four weeks that may be extended up to six weeks by mutual consent of the patients and the investigators.

Objectives:

1. To conduct Phase 2A to determine how tumor size, tumor tissue biomarkers, and the cancer stem cell markers, in head and neck squamous cell cancer patients are affected by the administration APG-157 pastilles using imaging and other clinical measurements.
2. To determine the degrees of response of each patient to APG-157 (considering patient's diagnosis/staging and local treatment) using proposed primary, secondary and exploratory endpoints.
3. The results from this study will be used to finalize the design of subsequent Phase 2B study (single arm for specific patient population and local treatment) to demonstrate statistically significant efficacy outcomes.

ELIGIBILITY:
Inclusion Criteria:

A. Biopsy proven oral cavity or oropharyngeal Squamous Cell Carcinoma.

B. Newly diagnosed, treatment naive Stage I, Stage II, Stage III or Stage IV HNSCC patients. Staging is done according to the International Union Against Cancer's (UICC) classification system for oral cancer. Acceptable TNM staging is T1-4, N0-2, M0.

C. Patients who are scheduled to receive the following therapy after APG-157 treatment.

1. Local Therapy with Curative Intent Surgery alone or surgery followed by radiation.
2. Therapy with Palliative Intent Radiation alone. Radiation with concurrent radiosensitizing chemotherapeutic agents only using QUAD-shot protocol. Radiosensitizing chemotherapeutic agents are limited to carboplatin or cetuximab.
3. Patients who refuse surgery or are unfit for any local therapy.

Exclusion Criteria:

A. Patients whose definitive, local treatment is available in less than four weeks from initial diagnosis. For example, some patients who are scheduled to receive chemo-radiation therapy as the local therapy with curative intent.

B. Pregnant women.

C. Prior Chemotherapy or radiation therapy within the last 8 weeks.

D. Patients with recurrent or metastatic cancer.

E. Tooth abscesses.

F. Bleeding gums or cracked teeth.

G. Patients who have had surgery of the oral cavity, teeth, or gums within the previous 8 weeks.

H. Patients who have had a fracture of the mandible or maxilla within the previous 8 weeks.

I. Inability to complete enrollment forms due to any mental status or language problems (e.g. dementia, head injury, overall illness).

J. Patients with other related diseases or the oral cavity or oropharynx, as determined to be significant by the PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Imaging to assess drug's ability to impact tumor size | Baseline to end of dosing is four weeks (extendable up to 6 weeks) of APG-157 dosing. Baseline is at time of diagnosis. End of dosing is day before surgery or start of other definitive therapy and/or radiation
  Change in Tumor Size from Baseline to end of dosing using MRI with or without contrast and PET/CT imaging.

SECONDARY OUTCOMES:
Biopsy | Baseline to end of dosing is four weeks (extendable up to 6 weeks) of APG-157 dosing. Baseline is at time of diagnosis. End of dosing is day before surgery or start of other definitive therapy and/or radiation
  Change in Immunohistochemistry profile (including the levels of tumor infiltrating lymphocytes TILs) of tumor biopsy from baseline to end of dosing.
Saliva Profile | Baseline to end of dosing is four weeks (extendable up to 6 weeks) of APG-157 dosing. Baseline is at time of diagnosis. End of dosing is day before surgery or start of other definitive therapy and/or radiation
  Change in cytokine levels (IL-1β , TNF-α, IL-8) and oral microbiome (phyla and genus level changes in microbial composition using 16s RNA sequencing) in saliva from baseline to end of dosing.
Cell-free RNA analyses of saliva and blood | Baseline to end of dosing is four weeks (extendable up to 6 weeks) of APG-157 dosing. Baseline is at time of diagnosis. End of dosing is day before surgery or start of other definitive therapy and/or radiation
  Change in cell-free RNA biomarkers in blood and saliva from baseline to end of dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Marilene B Wang, MD, Principal Investigator — VA Los Angeles/UCLA; Elizabeth Franzmann, MD, Principal Investigator — University of Miami Sylvester Comprehensive Cancer Center
Locations (2):
- United States (2):
  - VAGLAHS, West Los Angeles, Los Angeles, California
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida

IPD SHARING:
Plan to Share IPD: No